CLINICAL TRIAL: NCT04733092
Title: Prospective Study of the Safety and Efficacy of the Use of a Lipiodol Emulsion for the Embolization of Inflammatory Hypervascularizations Observed in Patients With Joint or Abarticular Knee Pain
Brief Title: Safety and Efficacy of a Lipiodol Emulsion for the Embolization of Hypervascularizations in Patients With Knee Pain (LipioJoint1)
Acronym: LipioJoint1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190891; 2020-002206-10 (EudraCT Number)
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
Keywords: Lipiodol; musculoskeletal disorders; embolization
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases | interventions — Ethiodized Oil; ioversol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization (Experimental): Embolization of the inflammatory hypervascularization with a lipiodol emulsion
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Drug: Lipiodol — Lipiodol in emulsion with contrast agent
  Other Names: Optiray

SUMMARY:
Knee osteoarthritis is a common cause of disability in patients who are often young and active. Surgery being an option only for the most severe cases, there is little alternative in case of failure of recommended medication. Inflammatory hypervascularization of the joint is a known source of pain. Temporary embolization of intra-arterial inflammatory hypervascularization has been used since 2012 with good results on pain relief to treat patients with musculoskeletal disorders that are resistant to conventional treatments. Lipiodol® has transient embolizing properties when in emulsion with a contrast agent. It has been used as an emulsion with chemotherapy for the treatment of metastases and primary intra-arterial liver cancer (chemo-embolization) for many years without serious side effects. We hypothesized that Lipiodol® in emulsion could serve as a temporary embolization agent for the treatment of inflammatory hypervascularization responsible for musculoskeletal disorders in humans.

DETAILED DESCRIPTION:
It is a Phase 1, Single-Arm, Open-label, Multicenter Interventional Prospective Study.

In order to ensure the best possible patient safety, a sequential inclusion of the first 6 patients is planned. Thus, the inclusion of each subsequent patient (patient 2-6) will only be considered after reviewing previously included patient safety data. Safety data after the inclusion of each patient (after a step-back of at least one week), as well as the cumulative review of previously included patient safety data, will be brought to the attention of all investigators involved in this research.

In addition, the following information will be transmitted to the Competent Authority without delay:

* a review of the safety and efficacy of the first 3 patients included with a step back for the last patient of at least one week after the administration of the experimental drug, as well as an argument as to the continuation of this research with regard to these data, with a discussion of the risks incurred in relation to the expected profit
* a review of the safety and effectiveness of the first 3 patients after the inclusion of the first 6 patients, as well as an argument as to the continuation of this research with regard to these data, with a discussion of the risks incurred compared to the expected benefit.

The patients will be embolized by the Interventional Radiology Department of the European Hospital Georges Pompidou (HEGP). Embolization will be performed by an experienced radiologist during a conventional hospitalization or a day hospitalization. A clinical follow-up will be carried out at 1 week, 1 month and 3 months after embolization by clinics and patient self-assessment (WOMAC, SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary inflammatory knee osteoarthritis of the target joint defined by a knee osteoarthritis according to the American College of Rheumatology (ACR) classification and a score ≥ 2 according to the classification of Kellgren and Lawrence
* Patient not eligible for surgery (or refusing surgery)
* Analog Visual Scale (VAS) pain ≥ 40 mm despite analgesic treatment for at least 3 months
* Failure or intolerance of treatment with NSAIDs and/or tramadol and/or acetaminophen, and/or failure or intolerance or patient refusing strong opioids medication (morphine, codeine)
* Failure or patient refusal of corticosteroid infiltration
* Patient who has signed an informed consent

Exclusion Criteria:

* Patient who is unable or unable to comply with the follow-up schedule
* Infiltration of target joint less than three months old
* Treated hyperthyroidism
* Traumatic injury, hemorrhage or bleeding less than 1 week old in the target joint
* Known arterial disease of the lower limbs stage ≥ 2 according to the classification of Leriche and Fontaine
* Known severe allergy to Lipiodol® and/or iodized contrast product
* Known severe kidney failure (creatinine clearance < 30 ml/min)
* Pregnant or breastfeeding woman
* Patient not affiliated with a French Medicare
* Patient benefiting from legal protection
* Participation in another interventional research

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events (SAE) | 1 month
  Number of SAE related to Embolization

SECONDARY OUTCOMES:
Immediate Technical success | Intraoperative
  Success of catheterization and embolization of target hypervascularization
Pain improvement 1 week after embolization | 1 week
  Analog Visual Scale score (0-100) comparison to baseline VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The Scale is rated from 0 to 100 (no pain to extremely severe pain)
Pain improvement 1 month after embolization | 1 month
  Analog Visual Scale score (0-100) comparison to baseline VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The Scale is rated from 0 to 100 (no pain to extremely severe pain)
Pain improvement 3 month after embolization | 3 months
  Analog Visual Scale score (0-100) comparison to baseline VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The Scale is rated from 0 to 100 (no pain to extremely severe pain)
Articular impotence improvement 1 week after embolization | 1 week
  Western Ontario and McMaster Universities Osteoarthritis Index score (0-96) comparison to baseline
Articular impotence improvement 1 month after embolization | 1 month
  Western Ontario and McMaster Universities Osteoarthritis Index score (0-96) comparison to baseline
Articular impotence improvement 3 month after embolization | 3 months
  Western Ontario and McMaster Universities Osteoarthritis Index score (0-96) comparison to baseline
Quality of life improvement 3 month after embolization | 3 months
  Short Form Health Survey (SF-36) score comparison to baseline SF-36 consists of eight scaled scores which are the weighted sums of the questions in their section, a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Pain medication improvement 1 week after embolization | 1 week
  Dose of analgesic medication compared to baseline (mg/24h)
Pain medication improvement 1 month after embolization | 1 month
  Dose of analgesic medication compared to baseline (mg/24h)
Pain medication improvement 3 month after embolization | 3 months
  Dose of analgesic medication compared to baseline (mg/24h)
Patient's satisfaction | 3 months
  Patient's satisfaction questionnaire : qualitative questionnaire with 5 ordered modalities (0 = no to 4 = yes)
Adverse Events (AE) | 3 months
  Number of AE related to embolization
Serious Adverse Events (SAE) | 3 months
  Number of SAE related to embolization

CONTACTS AND LOCATIONS:
Overall Officials: Marc MD Sapoval, PhD, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- Hôpital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: 2 years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contracting

REFERENCES:
- [Derived] Sapoval M, Querub C, Pereira H, Pellerin O, Boeken T, Di Gaeta A, Ahmar MA, Lefevre-Colau MM, Nguyen C, Daste C, Lacroix M, Laredo JD, Sabatier B, Martelli N, Chatellier G, Dean C, Rannou F. Genicular artery embolization for knee osteoarthritis: Results of the LipioJoint-1 trial. Diagn Interv Imaging. 2024 Apr;105(4):144-150. doi: 10.1016/j.diii.2023.12.003. Epub 2023 Dec 14. PMID 38102013